CLINICAL TRIAL: NCT06294028
Title: International Multicenter Project Comparing Radiofrequency Ablation Versus Implantable Defibrillator After Well-tolerated Ventricular Tachycardia in Ischemic Heart Disease with Minimally Impaired Ejection Fraction
Acronym: VIVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC31/21/0338
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Ischemic Heart Disease; Ventricular Tachycardia
Keywords: Ablation
MeSH Terms: conditions — Myocardial Ischemia; Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Implantation of an automatic defibrillator (Active Comparator): Implantation of an automatic defibrillator
  Interventions: Other: Adverse events collection; Other: Quality of life questionnaire EQ-5D-5L; Other: Medical-economic evaluation
- Percutaneous catheter ablation (Experimental): Percutaneous catheter ablation
  Interventions: Other: Adverse events collection; Other: Quality of life questionnaire EQ-5D-5L; Other: Medical-economic evaluation

INTERVENTIONS:
Other: Adverse events collection — Collection of deaths from any cause, hospitalizations or emergency consultations for any event related to ventricular arrhythmia or its treatment (recurrence of ventricular tachycardia or complication linked to the defibrillator or crossover from one group to another)
Other: Quality of life questionnaire EQ-5D-5L — Questionnaire on the patient's quality of life and health in 6 questions: on mobility, the person's autonomy, current activities, pain, anxiety. Answers range from "no problem" to "unable" and 5 possible answers to each question.
  The last question concerns the patient's health, the patient must rate his or her health on a scale of 0 to 100
Other: Medical-economic evaluation — Collection of expenses incurred by the care of patients in each arm will be collected over a period of 36 months.
  Direct medical and non-medical costs as well as costs related to absences from the workplace will be included in the analysis. Healthcare consumption will be collected using the National Health Data System (SNDS).

SUMMARY:
Evidence for the usefulness of the defibrillator in cases of preserved left ventricular ejection fraction and well-tolerated ventricular tachycardia (without cardiocirculatory arrest or syncope) is lacking, as no previous trials have included such patients. Additionally, sudden death in this particular population is low compared to other subgroups of patients with malignant ventricular arrhythmias.

On the other hand, numerous recent retrospective data show that ablation of ventricular tachycardia can reduce mortality, and also clearly reduces the number of recurrences in prospective studies.

Finally, a very low rate of sudden death was observed in a multicenter European retrospective study that we conducted, including patients with well-tolerated ventricular tachycardia in structural heart disease with minimally impaired ejection fraction and benefiting from ablation without implantation of defibrillator.

ELIGIBILITY:
Inclusion Criteria:

* ischemic heart disease with history of infarction - LVEF> 35% (measured by MRI)
* sustained monomorphic ventricular tachycardia - without history of syncope or cardiac arrest -
* having signed informed consent
* affiliated to a social security system

Exclusion Criteria:

* transient regressive cause of ventricular tachycardia
* recent myocardial infarction (<2 months)
* ventricular tachycardia by reentry from branch to branch
* serious conduction disturbances (with indication of stimulation)
* contraindication to the implantation of a defibrillator or to the performance of an ablation (life expectancy <1 year, relevant comorbidities)
* pregnancy
* age <18 years
* Patient under legal protection, guardianship or curatorship

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Monitoring for the occurrence of at least one serious event during the 36 months of follow-up | 36 months
  Monitoring of the occurrence of death from any cause, hospitalization or emergency consultation for any event related to ventricular arrhythmia or its treatment (recurrence of ventricular tachycardia or complication linked to the defibrillator or crossover from one group to another)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe MAURY, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Rangueil Hospital, Toulouse, France, France

IPD SHARING:
Plan to Share IPD: No